CLINICAL TRIAL: NCT03093792
Title: Effects of a Carbohydrate Restricted, High Protein, High Fat Diet on Weight Loss and Health Outcomes in Women Participating in the Curves Fitness and Weight Loss Program
Brief Title: Effects of Diet Manipulation on Women in the Curves Program
Acronym: Curves2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Curves International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB2013-0495FX
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Diet, Carbohydrate-Restricted
MeSH Terms: interventions — American Heart Association; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator): (no diet or exercise intervention)
  Interventions: Other: Control
- American Heart Association (Experimental): (AHA: 55% carbohydrate, 15% protein, 30% fat - diet plus exercise)
  Interventions: Other: American Heart Association plus exercise
- Curves Complete - I (Active Comparator): (CC - I: 30% carbohydrate, 45% protein, 25% fat - diet plus exercise)
  Interventions: Other: Curves Complete - I plus exercise
- Curves Complete - II (Active Comparator): (CC - II: 20% carbohydrate, 45% protein, 35% fat - diet plus exercise)
  Interventions: Other: Curves Complete - II plus exercise

INTERVENTIONS:
Other: Control
  Arms: Control
Other: American Heart Association plus exercise
  Arms: American Heart Association
Other: Curves Complete - I plus exercise
  Arms: Curves Complete - I
Other: Curves Complete - II plus exercise
  Arms: Curves Complete - II

SUMMARY:
The purpose of this study is to look at the effects of a carbohydrate restricted, high protein, high fat diet on weight loss and health outcomes in women participating in the Curves Fitness and Weight Loss Program.

DETAILED DESCRIPTION:
The purpose of this study is to determine if a carbohydrate restricted, high protein, high fat diet (20% carbohydrate, 45% protein, 35% fat; CC-II) promotes more favorable changes in weight loss and health outcomes compared to a traditional high carbohydrate, low protein, low fat diet (55% carbohydrate, 15% protein, 30% fat; AHA) and the Curves moderate carbohydrate restricted, high protein, and low fat diet (30% carbohydrate, 45% protein, 25% fat; CC-I).

ELIGIBILITY:
Inclusion Criteria:

* The participant is an apparently healthy female
* The participant is between the ages of 18 and 60

Exclusion Criteria:

* The participant is pregnant or nursing, or plans to become pregnant during the next 12 months or has been pregnant in the past 12 months
* The participant has uncontrolled metabolic disorder including known electrolyte abnormalities; heart disease, arrhythmias, diabetes, thyroid disease, or hypogonadism; a history of hypertension, hepatorenal, musculoskeletal, autoimmune, or neurological disease
* The participant is currently taking thyroid, hyperlipidemic, hypoglycemic, anti-hypertensive, or androgenic medications
* The participant has taken ergogenic levels of nutritional supplements that may affect muscle mass (e.g., creatine, HMB), anabolic/catabolic hormone levels (androstenedione, DHEA, etc.) or weight loss (e.g., ephedra, thermogenics, etc.) within the past three months
* The participant is willing to participate in a regular moderate exercise program

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The eligibility criteria were at the request of the study sponsor.
Enrollment: 86 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2015-05-01 (Actual)

PRIMARY OUTCOMES:
Effects of the Curves program on physical activity patterns | 24 weeks
Effects of the Curves program on body weight | 24 weeks
Effects of the Curves program on the hip/waist ratio | 24 weeks
Effects of the Curves program on Resting Energy Expenditure (REE) | 24 weeks
Effects of the Curves program on Blood Pressure (BP) | 24 weeks
Effects of the Curves program on Heart Rate (HR) | 24 weeks
Effects of the Curves program on body composition (DXA) | 24 weeks
Effects of the Curves program on Bioelectrical Impedance Analysis (BIA) | 24 weeks
Effects of the Curves program on a chemistry-15 blood panel | 24 weeks
Effects of the Curves program on a cell blood count (CBC) blood panel | 24 weeks
Effects of the Curves program on lipid panels | 24 weeks

SECONDARY OUTCOMES:
Effects of the Curves program on maximal cardiopulmonary capacity | 24 weeks
Effects of the Curves program on muscular strength through a 1 repetition maximum (1 RM) test | 24 weeks
Effects of the Curves program on muscular endurance through a maximal repetition test | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University

IPD SHARING:
Plan to Share IPD: No